CLINICAL TRIAL: NCT01724060
Title: The Effects of Current Treatments of Obesity on Food Preferences, Gut Hormones, Bile Acids and Hepatic Glucose Output in Humans.
Brief Title: Effects of Obesity Treatments on Food Preferences and Metabolism
Acronym: FPS
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: FPS
Record Dates: First submitted 2012-10-16; First posted 2012-11-09 (Estimated); Results first posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Obesity; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Human plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (8):
- Gastric bypass: Patients due for gastric bypass surgery
- Gastric banding: Patients due for gastric banding
- Sleeve gastrectomy: Patients due for sleeve gastrectomy
- Endobarrier: Patients due to undergo endoscopic Endobarrier insertion
- Exenatide: Patients due to be commenced on Exenatide
- Liraglutide: Patients due to be commenced on Liraglutide
- Lifestyle: Patients due to be commenced on a lifestyle intervention programme
- Elective surgery or endoscopy: Patients due to have non bariatric surgery (i.e. cholecystectomy) or an elective diagnostic endoscopy

SUMMARY:
Obesity and Type 2 Diabetes Mellitus are major health problems which are becoming a burden both for patients and health systems alike. The surgical and medical treatments available for these conditions have improved significantly in the last two decades. The investigators do not however know how these treatments compare to each other and how they act in the body to cause weight loss and diabetes improvements. The studies of this experiment are complementary to each other. They aim to answer related questions and will allow us to study how these treatments work and eventually develop safer and more effective therapies for obesity and diabetes.

DETAILED DESCRIPTION:
The objective of this study is to investigate the effects of obesity surgical procedures and incretin therapies on food preferences, satiety, gut hormones, bile acids and hepatic glucose output in overweight and obese patients.

As part of routine care these patients will be seen by a dietician/diabetes specialist nurse (DSN) before and after intervention. Patients will be asked to prospectively complete food diaries on three consecutive days which are representative of their usual dietary intake. The first food diary will be completed three months to two weeks pre intervention. Another four food diaries will be completed post intervention: at one, three months, 6 months and one year. Total energy intake and macronutrient composition comparisons pre and post intervention will form the basis of our analysis.

20 patients in each group will undergo more detailed measurements of food intake, hunger, satiety, gut hormones and bile acids. The research protocol will be the similar to that previously published by the Department of Metabolic Medicine, Imperial College, London. Participants will be fasted for 12 hours overnight and will attend for the study on 5 occasions. On each occasion venous blood samples will be taken and visual analogue scores will be measured over a 3 hour period using previously published methodology Samples or sample containers will be anonymised before collection but will be traceable back to the individual patients. Urine will be collected once. A qualified medical doctor will insert a venepuncture cannula into the arm of the patient and 5ml blood will be withdrawn at baseline, 15, 30, 60, 90, 120, 150 and 180 minutes following ingestion of a standard 400kcal meal as below.

Ten patients in each group (different from those taking part in the meal studies) will undergo measurements of hepatic glucose output/insulin resistance through euglycaemic hyperinsulinaemic clamps (Metabolic Study). To ensure that acute caloric restriction does not affect insulin sensitivity, patients will be on a low calorie liquid diet for 4-14 days and 3-7 days after intervention to ensure that their weight is stable throughout the study. This diet is nutritious and contains all appropriate macronutrients. Such diets are frequently used as part of pre-obesity interventions to reduce weight and risk. Patients will provide the investigators with a detailed food diary of their food consumption for this period.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with overweight and/or obesity (BMI ≥30 Kg/m2) who are eligible for obesity treatment based on NICE guidance or that are having non bariatric surgery or endoscopy.

Exclusion Criteria:

* None

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients from the community or hospital care
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2012-09; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carel W le Roux, MRCP PhD, Principal Investigator — Imperial College London
Locations (2):
- United Kingdom (2):
  - Royal Surrey County Hospital, Guildford
  - Imperial Weight Centre, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were no pre assignments requirements
Period: Overall Study
Arm/Group | Gastric Bypass | Gastric Banding | Sleeve Gastrectomy | Endobarrier | Exenatide | Liraglutide | Lifestyle | Elective Surgery or Endoscopy
Started | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients attending obesity clinic from living in a multinational city such as London.
Groups:
- Total: Total of all reporting groups
Arm/Group | Gastric Bypass | Gastric Banding | Sleeve Gastrectomy | Endobarrier | Exenatide | Liraglutide | Lifestyle | Elective Surgery or Endoscopy | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 80
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: year] | 42 (12) | 40 (14) | 44 (9) | 43 (7) | 44 (8) | 41 (7) | 43 (13) | 40 (15) | 42 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 6 | 4 | 7 | 6 | 3 | 5 | 41
  Male | 5 | 5 | 4 | 6 | 3 | 4 | 7 | 5 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 80
Region of Enrollment [Number; unit: participants]
  United Kingdom | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 80
Food Intake [Mean (Standard Deviation); unit: kcal] | 1505 (205) | 1490 (218) | 1482 (162) | 1511 (197) | 1503 (222) | 1420 (183) | 1471 (193) | 1453 (211) | 1503 (198)

OUTCOME MEASURES:

1. Primary Outcome: Change in Energy Intake From Baseline
Description: The difference in total calories consumption between baseline and 12 months
Time Frame: Change at 12 months
Population: Patients that had specific obesity interventions.
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Gastric Bypass | Gastric Banding | Sleeve Gastrectomy | Endobarrier | Exenatide | Liraglutide | Lifestyle | Elective Surgery or Endoscopy
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
kcal | 500 (55) | 310 (76) | 482 (69) | 5 (105) | 27 (92) | 103 (74) | 11 (129) | 15 (114)

2. Secondary Outcome: Change in Appetite Ratings From Baseline
Description: Visual Analogues difference between baseline and follow up
Time Frame: Change 12 months
Reporting Status: Not Posted

3. Secondary Outcome: Change in Metabolites From Baseline
Description: Blood samples difference between baseline and follow up
Time Frame: Change at 12 months
Reporting Status: Not Posted

4. Secondary Outcome: Change in Hepatic Insulin Resistance From Baseline
Description: Insulin clamps difference between baseline and follow up
Time Frame: Change at 1 week after intervention
Reporting Status: Not Posted

5. Secondary Outcome: Change in Macronutrient Composition From Baseline
Description: Macronutrients difference between baseline and follow up
Time Frame: Change at 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Description: No difference
Groups:
- Elective Surgery or Endoscopy: Patients due to have non bariatric surgery (i.e. cholecystectomy) or an elective diagnostic endoscopy. No adverse events recorded.
Arm/Group | Gastric Bypass | Gastric Banding | Sleeve Gastrectomy | EndoBarrier | Exenatide | Liraglutide | Lifestyle | Elective Surgery or Endoscopy
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
The study was limited by different treatment modalities being compared such as endobarrier, gastric bypass and medication

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-06-12): https://cdn.clinicaltrials.gov/large-docs/60/NCT01724060/Prot_SAP_000.pdf